CLINICAL TRIAL: NCT06212726
Title: Evaluation of Return-to-learn Concussion Management Coordination and Social Determinants of Health on Patient-centered Outcomes
Brief Title: RTL Concussion Communication
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators left the institution
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202301378
Record Dates: First submitted 2023-09-19; First posted 2024-01-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Concussion, Mild; Post Concussion Symptoms; Cognitive Impairments; Cognitive Impairments, Mild; Multidisciplinary Care Team; Team Nursing; Sports Injuries in Children; Learning Disturbance
Keywords: concussion; Post-concussion syndrome; return to learn; return to school; concussion management; multidisciplinary care team; Interdisciplinary team; Implementation science; communication
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Cognitive Dysfunction; Learning Disabilities; Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InjureFree Concussion Communication Tool (Experimental): During the second phase of this trial, participants assigned to the experimental group (Buchholz and Gainesville High Schools) will receive the current standard of care for return to learn following SRRC with the addition of InjureFree, a wed-based injury tracking and communication tool. InjureFree will serve as a centralized area for concussion management team members to communicate and document participant progress with the return to learn program.
  Interventions: Behavioral: InjureFree
- Control (No Intervention): During the second phase of this trial, participants assigned to the control group (Newberry, Santa Fe and Eastside High Schools) Will not receive any intervention other than the current standard of care for return to learn following SRRC currently in place.

INTERVENTIONS:
Behavioral: InjureFree — The InjureFree software is a commercialized injury incident management platform for organizations working in sports and athlete care and is focused on providing administrators and caregivers' technology to enhance coordination of care. InjureFree will be utilized to track concussion management and communication following SRRC at Buchholz and Gainesville High Schools. This will not modify the current standard of practice for healthcare delivery, it will only modify the communication between members of the concussion management team
  Arms: InjureFree Concussion Communication Tool

SUMMARY:
This study is aimed at improving health outcomes for adolescents who sustain sport and recreation related concussions (SRRC) by enhancing Return to Learn (RTL). The study will conduct a quasi-experimental school-based 2 phase study involving 200 students with SRRC. The first phase will be descriptive to evaluate current standards (n=50). Phase 2 will compare students whod receive either standard of care RTL (n=75) or RTL augmented by a communication tool (RTC+; n=75).

DETAILED DESCRIPTION:
Up to 3.8 million secondary school students are diagnosed with a sport and recreation related concussion (SRRC) annually in the U.S., which can have a detrimental impact on educational attainment, a social determinant of health (SDOH) that is linked with college admission and graduation, employment, income status and social class. This research will address this significant public health problem by gaining a deeper understanding of the relationships among SRRC and SDOH and examine the impact of concussion management team communication on return to learn (RTL) outcomes for students following an SRRC. This research has significant potential to improve RTL outcomes of secondary school students and may provide evidence to support policy-level changes to reduce disparities in SRRC management, especially among low-resource school districts.

The three research aims of this study will proceed as follows:

Aim 1 will examine the relationships among SDOH, SRRC-related symptoms, and RTL milestones among a diverse population of adolescents and young adult secondary school students following SRRC. This aim will be achieved by enrolling and tracking secondary school students who sustain an SRRC over a 12-month period.

Aim 2 will compare RTL milestones among secondary school students following SRRC who are managed by an interdisciplinary concussion management team that uses standard or care plus a communication tool intervention or only standard of care for the RTL process.

Aim 3 will examine differential RTL outcomes between groups (standard of care plus a communication tool intervention vs. only standard of care) based on SDOH, sex as a biological variable, and pre-injury health status among secondary school students following SRRC.

The study aims to reduce disparities in timely management of SRRC during the process of RTL, achievement of RTL milestones and improvement of SRRC-related symptoms in the context of SDOH.

ELIGIBILITY:
Inclusion Criteria:

* Student: enrolled in Alachua County Public Secondary Schools who are age 14 or older and have sustained a new SRRC and voluntarily enrolled in the OSMI (Orthopaedic Sports Medicine Institute) concussion management program
* Parent: primary point of contact for the assenting student verified through the school

Exclusion Criteria:

* Student: Age 13 or younger, Not enrolled in Alachua County Public Schools, Did not sustain SRRC during school year
* Parent: not a verified point of contact for the assenting student

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Participant self-efficacy in concussion symptom management | 1 month
  Participant will demonstrate increased ability in self-management of post-concussion symptoms. To measures self efficacy, the research team will utilize a 10-item scale with answers on a likert scale from 1-10 with 1 being not at all confident and 10 being completely confident. Examples of items are: How confident are you that you can manage your concussion symptoms with the instructions provided by the Concussion Management Team (CMT)? How confident are you that you can manage your return to the classroom with the instructions provided by the CMT? How confident are you that you can judge when the changes in your concussion symptoms means you should visit a doctor? How confident are you that you can exercise without making concussion symptoms worse? How confident are you that you can keep the symptoms of your concussion from interfering with the things you want to do?
Communication satisfaction | 1 month
  Participant will express level of satisfaction with concussion management team (CMT) communication and care delivery throughout the return to learn (RTL) process. RTL communication satisfaction will be measured with a series of questions. The questions will consist of 5 items asking about levels of satisfaction with care coordination, availability of providers and CMT members, education on SRRC provided, understanding of RTL process and frequency of communication from CMT members during RTL. A 4-point Likert scale will be used ranging from not at all satisfied to very satisfied.

SECONDARY OUTCOMES:
Post concussion symptom reduction | 1 month
  Participant will experience a decreased symptom burden as evidenced by scores utilizing the Post-Concussion Symptom Scale (PCSS). The PCSS is a widely used tool for assessing post-concussion symptoms. It measures various physical, cognitive, and emotional symptoms that individuals may experience following a concussion. Participants indicate symptom severity on a scale from 0-6 with zero being no symptoms and six being severe symptoms. Possible scores range from 0 to 132 with higher scores indicating a more severe burden of symptoms.

IPD SHARING:
Plan to Share IPD: No
IDP will be made available to other researchers upon request. Only de-identified information will be made available.